CLINICAL TRIAL: NCT01408901
Title: PROgenitor Cell Release Plus Exercise to Improve functionaL Performance in PAD: The PROPEL Study
Brief Title: Treadmill Exercise and GM-CSF Study to Improving Functioning in Peripheral Artery Disease (PAD)
Acronym: PROPEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary McDermott, Professor of Medicine and Preventive Medicine at Northwestern University Feinberg School of Medicine, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00049675; R01HL107510 (NIH)
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Results first posted 2019-12-10 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; granulocyte macrophage colony stimulating factor; PAD; GM-CSF; sargramostim; leukine; treadmill exercise
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A: GM-CSF + supervised treadmill exercise therapy (Experimental)
  Interventions: Behavioral: Supervised Treadmill Exercise Therapy; Drug: granulocyte macrophage colony stimulating factor (GM-CSF)
- B: GM-CSF + attention control group (Active Comparator)
  Interventions: Other: Health education sessions (Control); Drug: granulocyte macrophage colony stimulating factor (GM-CSF)
- C: placebo + supervised exercise therapy (Active Comparator)
  Interventions: Behavioral: Supervised Treadmill Exercise Therapy
- D: placebo + attention control group (Placebo Comparator)
  Interventions: Other: Health education sessions (Control)

INTERVENTIONS:
Behavioral: Supervised Treadmill Exercise Therapy — Exercise intervention will be delivered three times weekly for 26 weeks. In the first week, participants will be asked to exercise 15 minutes per session (excluding rest periods). Walking exercise duration will be increased to 25 minutes minutes per session during week 2. Week 3 and 4 sessions will also be 25 minutes long, but the intensity will be increased either to produce leg symptoms or at a target rate of perceived exertion (RPE)of 12-14 on the Borg's 6-20 scale. For weeks 5-8, walking duration will be increased to 40 to 50 minutes while maintaining intensity. For weeks 9-26, exercise duration will continue to be 40 to 50 minutes but we will increase intensity up to a maximum of 4.0 miles per hour at 10% grade.
  Other Names: treadmill exercise
  Arms: A: GM-CSF + supervised treadmill exercise therapy; C: placebo + supervised exercise therapy
Other: Health education sessions (Control) — Participants randomized to the attention control group will attend weekly one-hour educational sessions at Northwestern University for six months. These educational sessions are on topics of interest to the typical PAD patient and are led by physicians and other health care workers. Topics include Medicare Part D, nutritional supplements, C-reactive protein, and hypertension. Sessions do not include information about exercise.
  Other Names: attention control group
  Arms: B: GM-CSF + attention control group; D: placebo + attention control group
Drug: granulocyte macrophage colony stimulating factor (GM-CSF) — The dose of GM-CSF will be 250 ug/M^2 subcutaneously three times weekly for two weeks.
  Other Names: sargramostim; leukine
  Arms: A: GM-CSF + supervised treadmill exercise therapy; B: GM-CSF + attention control group

SUMMARY:
The PROPEL study will test the hypothesis that GM-CSF combined with supervised treadmill exercise will significantly improve functional performance in patients with PAD more than GM-CSF alone or supervised treadmill exercise alone. In addition to identifying novel therapeutic options for patients with PAD, the current proposal is expected to identify mechanisms by which functional impairment is improved in patients with PAD.

DETAILED DESCRIPTION:
Eight million men and women in the United States have lower extremity peripheral arterial disease (PAD). PAD is expected to be increasingly common as the population survives longer with chronic disease. Patients with PAD have greater functional impairment and faster functional decline compared to those without PAD. However, currently there are only two FDA approved medications for improving functional performance in patients with PAD. Furthermore, these FDA approved medications are only modestly beneficial for improving walking performance in patients with PAD.

Preliminary evidence suggests that increasing circulating levels of CD34+ cells with granulocyte macrophage colony stimulating factor (GM-CSF) or other therapies may improve walking performance in patients with PAD. However, results of small clinical trials testing the ability of GM-CSF to improve walking performance in patients with PAD are mixed. The association of GM-CSF with improved walking performance in PAD is not definitively established. Preliminary data also suggest that lower extremity ischemia, induced during walking exercise, may increase circulating CD34+ cell levels, enhance homing of CD34+ cells to ischemic sites, and augment the ability of GMCSF to improve walking performance in PAD. However, it is currently unknown whether the combination of GM-CSF and supervised treadmill exercise significantly improve functional performance more than either therapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with an ankle brachial index (ABI) ≤ 0.90 will be eligible for participation.
2. Participants with an ABI > 0.90 but ≤ 1.00 who experience a 20% drop in ankle pressure after the heel-rise exercise will be eligible.
3. Participants with an ABI > 0.90 who have medical record evidence of prior lower extremity revascularization and experience a 20% drop in ankle pressure after the heel-rise exercise will be eligible for inclusion.
4. Participants with an ABI > 0.90 who have medical record evidence of a non-invasive vascular laboratory test result consistent with PAD. Note that a screen-positive test from Lifeline Screening is not sufficient for inclusion in the study.

Exclusion Criteria:

The following exclusion criteria will be initially assessed by telephone:

1. Below or above-knee amputation.
2. Wheelchair confinement.
3. Use of a walking aid other than a cane (i.e. people using walkers).
4. Non-English speaking.
5. Significant hearing impairment.
6. Significant visual impairment.
7. Diagnosis of Parkinson's disease.
8. Inability to return to the medical center at the required visit frequency (three times per week).
9. > Class II New York Heart Association heart failure or angina (symptoms at rest or with minimal exertion).
10. Any increase in angina pectoris symptoms during the previous 6 months or angina at rest.
11. Foot ulcer. (Participants with a foot ulcer will be excluded by telephone and/or during a baseline study visit).
12. Lower extremity revascularization in the last three months or major orthopedic surgery during the previous three months.
13. Myocardial infarction, stroke, or coronary artery bypass grafting during the previous 3 months.
14. Major medical illnesses including end stage renal disease requiring dialysis and chronic lung disease requiring oxygen, since these individuals may not be able to adhere to study requirements. Participants who only use oxygen at night may still qualify.
15. Potential participants who have received G-CSF, GM-CSF, or erythropoietin within the past year will be excluded because these interventions may influence study outcomes independently of the interventions.
16. Pre-menopausal women will be excluded because cyclic estrogen changes can influence progenitor cell levels.
17. Potential participants with diabetes and documented proliferative retinopathy will be excluded because GM-CSF may exacerbate this condition.
18. Potential participants with a history of myeloid malignancy will be excluded because GM-CSF may exacerbate these conditions.
19. Potential participants who have been treated for late stage cancer during the past three years, since GM-CSF may theoretically activate quiescent cancer cells.
20. Planned lower extremity revascularization within the next 6 months.
21. Current participation in another clinical trial. If a participant recently completed a clinical trial, at least three months must have passed before they can be considered for the PROPEL Trial. However, for a clinical trial of stem cell or gene therapy intervention, potential participants will be potentially eligible immediately after the final study visit of the stem cell or gene therapy clinical trial, so long as at least six months has passed since the participant received their final treatment in the stem cell or gene therapy intervention.
22. Walking for exercise at a level comparable to that targeted in our intervention.
23. Current participation in or completion of a cardiac rehabilitation program within the last six months.

    The following exclusion criteria will be assessed at the time of the study visit or later:
24. Severe aortic stenosis identified by physical exam at the study visit.
25. Critical limb ischemia identified by physical exam at the study visit.
26. Coronary ischemia during exercise, defined as ST segment depression > 1 mm during the baseline exercise treadmill test, with or without associated chest discomfort, without a perfusion stress test demonstrating no reversible ischemia within the previous 3 months.
27. Left-bundle branch block or significant ST-T wave changes on the baseline ECG without a perfusion stress test demonstrating no reversible ischemia within the previous 3 months.
28. Stopping during the treadmill stress test for shortness of breath, chest pain, hip pain, knee pain, or another symptom that may not represent ischemic leg pain.
29. Stopping during the six-minute walk test for symptoms other than ischemic leg symptoms.
30. Foot ulcer identified at the study visit.
31. Mini-Mental Status Examination (MMSE) score < 23 or disabling psychiatric disease.
32. Failure to complete a study run-in period.
33. Walking impairment due to a cause other than PAD.

In addition to the exclusion criteria listed above, individuals thought to be poorly suited to the intervention (i.e. not a good fit) can be excluded at the discretion of the principal investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2011-09; Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary M McDermott, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Domanchuk K, Ferrucci L, Guralnik JM, Criqui MH, Tian L, Liu K, Losordo D, Stein J, Green D, Kibbe M, Zhao L, Annex B, Perlman H, Lloyd-Jones D, Pearce W, Taylor D, McDermott MM. Progenitor cell release plus exercise to improve functional performance in peripheral artery disease: the PROPEL Study. Contemp Clin Trials. 2013 Nov;36(2):502-9. doi: 10.1016/j.cct.2013.09.011. Epub 2013 Sep 27. PMID 24080099
- [Background] Saber R, Liu K, Ferrucci L, Criqui MH, Zhao L, Tian L, Guralnik JM, Liao Y, Domanchuk K, Kibbe MR, Green D, Perlman H, McDermott MM. Ischemia-related changes in circulating stem and progenitor cells and associated clinical characteristics in peripheral artery disease. Vasc Med. 2015 Dec;20(6):534-43. doi: 10.1177/1358863X15600255. Epub 2015 Aug 31. PMID 26324152
- [Background] McDermott MM, Guralnik JM, Criqui MH, Liu K, Kibbe MR, Ferrucci L. Six-minute walk is a better outcome measure than treadmill walking tests in therapeutic trials of patients with peripheral artery disease. Circulation. 2014 Jul 1;130(1):61-8. doi: 10.1161/CIRCULATIONAHA.114.007002. No abstract available. PMID 24982117
- [Background] McDermott MM. Lower extremity manifestations of peripheral artery disease: the pathophysiologic and functional implications of leg ischemia. Circ Res. 2015 Apr 24;116(9):1540-50. doi: 10.1161/CIRCRESAHA.114.303517. PMID 25908727
- [Result] McDermott MM, Ferrucci L, Tian L, Guralnik JM, Lloyd-Jones D, Kibbe MR, Polonsky TS, Domanchuk K, Stein JH, Zhao L, Taylor D, Skelly C, Pearce W, Perlman H, McCarthy W, Li L, Gao Y, Sufit R, Bloomfield CL, Criqui MH. Effect of Granulocyte-Macrophage Colony-Stimulating Factor With or Without Supervised Exercise on Walking Performance in Patients With Peripheral Artery Disease: The PROPEL Randomized Clinical Trial. JAMA. 2017 Dec 5;318(21):2089-2098. doi: 10.1001/jama.2017.17437. PMID 29141087
- [Derived] McDermott MM, Zhang D, Zhao L, Polonsky T, Ferrucci L, Ho KJ, Kibbe MR, Guralnik JM, Criqui MH, Tian L. Duration of Supervised Exercise Necessary for Meaningful Improvement in Peripheral Artery Disease. J Am Heart Assoc. 2025 Sep 16;14(18):e040058. doi: 10.1161/JAHA.124.040058. Epub 2025 Sep 5. PMID 40913279
- [Derived] Hammond MM, Tian L, Zhao L, Zhang D, McDermott MM. Attendance at Supervised Exercise Sessions and Walking Outcomes in Peripheral Artery Disease: Results From 2 Randomized Clinical Trials. J Am Heart Assoc. 2022 Dec 20;11(24):e026136. doi: 10.1161/JAHA.122.026136. Epub 2022 Dec 19. PMID 36533626
- [Derived] McDermott MM, Tian L, Criqui MH, Ferrucci L, Greenland P, Guralnik JM, Kibbe MR, Li L, Sufit R, Zhao L, Polonsky TS. Perceived Versus Objective Change in Walking Ability in Peripheral Artery Disease: Results from 3 Randomized Clinical Trials of Exercise Therapy. J Am Heart Assoc. 2021 Jun 15;10(12):e017609. doi: 10.1161/JAHA.120.017609. Epub 2021 Jun 2. PMID 34075780
- [Derived] Patel K, Polonsky TS, Kibbe MR, Guralnik JM, Tian L, Ferrucci L, Criqui MH, Sufit R, Leeuwenburgh C, Zhang D, Zhao L, McDermott MM. Clinical characteristics and response to supervised exercise therapy of people with lower extremity peripheral artery disease. J Vasc Surg. 2021 Feb;73(2):608-625. doi: 10.1016/j.jvs.2020.04.498. Epub 2020 May 19. PMID 32416309
- [Derived] Kosmac K, Gonzalez-Freire M, McDermott MM, White SH, Walton RG, Sufit RL, Tian L, Li L, Kibbe MR, Criqui MH, Guralnik JM, S Polonsky T, Leeuwenburgh C, Ferrucci L, Peterson CA. Correlations of Calf Muscle Macrophage Content With Muscle Properties and Walking Performance in Peripheral Artery Disease. J Am Heart Assoc. 2020 May 18;9(10):e015929. doi: 10.1161/JAHA.118.015929. Epub 2020 May 9. PMID 32390569
- [Derived] McDermott MM, Polonsky TS, Guralnik JM, Ferrucci L, Tian L, Zhao L, Stein J, Domanchuk K, Criqui MH, Taylor DA, Li L, Kibbe MR. Racial Differences in the Effect of Granulocyte Macrophage Colony-Stimulating Factor on Improved Walking Distance in Peripheral Artery Disease: The PROPEL Randomized Clinical Trial. J Am Heart Assoc. 2019 Jan 22;8(2):e011001. doi: 10.1161/JAHA.118.011001. PMID 30661439
- [Derived] Berroug J, Korcarz CE, Mitchell CK, Weber JM, Tian L, McDermott MM, Stein JH. Brachial artery intima-media thickness and grayscale texture changes in patients with peripheral artery disease receiving supervised exercise training in the PROPEL randomized clinical trial. Vasc Med. 2019 Feb;24(1):12-22. doi: 10.1177/1358863X18804050. Epub 2018 Nov 12. PMID 30418100

RESULTS

PARTICIPANT FLOW:
Period: 6-Week Follow-Up
Arm/Group | A: GM-CSF + Supervised Treadmill Exercise Therapy | B: GM-CSF + Attention Control Group | C: Placebo + Supervised Exercise Therapy | D: Placebo + Attention Control Group
Started | 53 | 53 | 53 | 51
Completed | 50 | 51 | 50 | 47
Not Completed | 3 | 2 | 3 | 4
Not completed — Lost to Follow-up | 2 | 1 | 3 | 2
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Cancelled visit | 0 | 1 | 0 | 2
Period: 12-Week Follow-Up (Primary Endpoint)
Arm/Group | A: GM-CSF + Supervised Treadmill Exercise Therapy | B: GM-CSF + Attention Control Group | C: Placebo + Supervised Exercise Therapy | D: Placebo + Attention Control Group
Started | 50 | 52 | 50 | 49
Completed | 49 | 50 | 50 | 46
Not Completed | 1 | 2 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Cancelled visit | 0 | 2 | 0 | 1
Period: 26-Week Follow-Up
Arm/Group | A: GM-CSF + Supervised Treadmill Exercise Therapy | B: GM-CSF + Attention Control Group | C: Placebo + Supervised Exercise Therapy | D: Placebo + Attention Control Group
Started | 49 | 52 | 50 | 47
Completed | 48 | 50 | 50 | 46
Not Completed | 1 | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: GM-CSF + Supervised Treadmill Exercise Therapy | B: GM-CSF + Attention Control Group | C: Placebo + Supervised Exercise Therapy | D: Placebo + Attention Control Group | Total
Number analyzed (Participants) | 53 | 53 | 53 | 51 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (9.5) | 67.9 (7.5) | 67.5 (8.7) | 66.0 (8.6) | 67.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 23 | 20 | 82
  Male | 33 | 34 | 30 | 31 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 3 | 9
  Not Hispanic or Latino | 51 | 51 | 51 | 48 | 201
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1 | 2
  Black or African American | 35 | 35 | 33 | 38 | 141
  White | 18 | 16 | 19 | 11 | 64
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ankle-brachial index (ABI) [Mean (Standard Deviation); unit: ratio] — The ABI measures systolic blood pressures in the right brachial, dorsalis pedis, and posterior tibial arteries and left dorsalis pedis, posterior tibial, and brachial arteries. Measurements are repeated. The ABI iscalculated by dividing mean pressures in each leg by the mean of the 4 brachial pressures.
  ratio | 0.70 (0.20) | 0.71 (0.17) | 0.69 (0.19) | 0.69 (0.19) | 0.70 (0.19)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.7 (6.5) | 30.7 (6.9) | 31.7 (6.0) | 29.9 (6.8) | 30.5 (6.6)
Six-minute walk distance [Mean (Standard Deviation); unit: meters] | 336.4 (109.5) | 339.8 (101.0) | 338.7 (95.6) | 339.1 (92.0) | 338.5 (99.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Six-Minute Walk Performance at 12-week Follow-up
Description: In the six-minute walk, participants walk back and forth along a 100-ft hallway for six minutes after standardized instructions to complete as many laps as possible. Distance covered in six minutes is recorded.
Time Frame: change from baseline to week 12
Population: Data were imputed for participants who were lost to follow-up or who canceled the visit. Variables used for imputation were age, ankle brachial index, body mass index, sex, race, smoking status, baseline outcome values, leg symptoms, and comorbidities. SAS procedure MI was used to obtain 20 imputed data sets.
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | A: GM-CSF + Supervised Treadmill Exercise Therapy | B: GM-CSF + Attention Control Group | C: Placebo + Supervised Exercise Therapy | D: Placebo + Attention Control Group
Number analyzed (Participants) | 51 | 53 | 53 | 51
meters | 22.2 [5.4 to 39.0] | -6.4 [-23.0 to 10.1] | 28.5 [11.7 to 45.4] | -5.0 [-22.3 to 12.2]
Statistical Analysis 1: Comparison: A: GM-CSF + Supervised Treadmill Exercise Therapy vs B: GM-CSF + Attention Control Group; Test type: Superiority; p = 0.052, t-test, 2 sided — The P value is a Hochberg-adjusted P value; Mean Difference (Final Values) = 28.7, 95% CI 2-sided [5.1 to 52.3]
Statistical Analysis 2: Comparison: A: GM-CSF + Supervised Treadmill Exercise Therapy vs C: Placebo + Supervised Exercise Therapy; Test type: Superiority; p = 0.91, t-test, 2 sided — The P value is a Hochberg-adjusted P value; Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-30.2 to 17.6]
Statistical Analysis 3: Comparison: B: GM-CSF + Attention Control Group vs D: Placebo + Attention Control Group; Test type: Superiority; p = 0.91, t-test, 2 sided — The P value is a Hochberg-adjusted P value; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-25.2 to 22.4]
Statistical Analysis 4: Comparison: C: Placebo + Supervised Exercise Therapy vs D: Placebo + Attention Control Group; Test type: Superiority; p = 0.02, t-test, 2 sided — The P value is a Hochberg-adjusted P value; Mean Difference (Final Values) = 33.6, 95% CI 2-sided [9.4 to 57.7]

2. Secondary Outcome: Change in Brachial Artery Flow-mediated Dilation (FMD) at 12-week Follow-up
Description: The brachial artery is imaged 5 to 9 cm above the antecubital fossa using a linear array vascular ultrasound transducer. Three video sequences are obtained. The first verifies the location and baseline hemodynamic state of the brachial artery. The second begins 20 seconds before cuff inflation and continues for 10 seconds after inflation. The third begins 15 seconds before cuff release and continues for 90 seconds after deflation. Brachial artery FMD is calculated as the percent change in brachial artery diameter at 60 seconds and at 90 seconds after the release of the cuff.
Time Frame: change from baseline to week 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | A: GM-CSF + Supervised Treadmill Exercise Therapy | B: GM-CSF + Attention Control Group | C: Placebo + Supervised Exercise Therapy | D: Placebo + Attention Control Group
Number analyzed (Participants) | 51 | 53 | 53 | 51
percent change | -0.37 [-2.50 to 1.28] | 0.10 [-1.49 to 1.18] | 0.14 [-1.53 to 1.50] | -0.72 [-2.02 to 1.64]
Statistical Analysis 1: Comparison: A: GM-CSF + Supervised Treadmill Exercise Therapy vs B: GM-CSF + Attention Control Group; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney) — The P value is a Hochberg-adjusted P value; Hodges-Lehmann estimator = -0.61, 95% CI 2-sided [-1.67 to 0.44]
Statistical Analysis 2: Comparison: A: GM-CSF + Supervised Treadmill Exercise Therapy vs C: Placebo + Supervised Exercise Therapy; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney) — The P value is a Hochberg-adjusted P value; Hodges-Lehmann estimator = -0.67, 95% CI 2-sided [-1.84 to 0.51]
Statistical Analysis 3: Comparison: B: GM-CSF + Attention Control Group vs D: Placebo + Attention Control Group; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney) — The P value is a Hochberg-adjusted P value; Hodges-Lehmann estimator = 0.36, 95% CI 2-sided [-0.66 to 1.38]
Statistical Analysis 4: Comparison: C: Placebo + Supervised Exercise Therapy vs D: Placebo + Attention Control Group; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney) — The P value is a Hochberg-adjusted P value; Hodges-Lehmann estimator = 0.48, 95% CI 2-sided [-0.64 to 1.59]

3. Secondary Outcome: Change in Maximal Treadmill Walking Time at 12-week Follow-up
Description: The Gardner graded treadmill exercise test is the standard, accepted treadmill protocol for measuring change in maximal treadmill walking time in response to interventions among PAD participants. In the Gardner exercise protocol, speed is maintained at 2.0 miles per hour (mph) and treadmill grade increases by 2.0% every two minutes. If patients cannot begin walking at 2.0 mph, treadmill speed is started at 0.50 mph and increased by 0.50 mph every 2 minutes until the participant reaches 2.0 mph, after which the treadmill grade is increased every two minutes.
Time Frame: change from baseline to week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | A: GM-CSF + Supervised Treadmill Exercise Therapy | B: GM-CSF + Attention Control Group | C: Placebo + Supervised Exercise Therapy | D: Placebo + Attention Control Group
Number analyzed (Participants) | 51 | 53 | 53 | 51
minutes | 3.5 [2.5 to 4.5] | -0.1 [-1.1 to 0.9] | 4.2 [3.2 to 5.2] | 0.5 [-0.6 to 1.6]
Statistical Analysis 1: Comparison: A: GM-CSF + Supervised Treadmill Exercise Therapy vs B: GM-CSF + Attention Control Group; Test type: Superiority; p < 0.01, t-test, 2 sided — The P value is a Hochberg-adjusted P value; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [2.1 to 5.0]
Statistical Analysis 2: Comparison: A: GM-CSF + Supervised Treadmill Exercise Therapy vs C: Placebo + Supervised Exercise Therapy; Test type: Superiority; p = 0.44, t-test, 2 sided — The P value is a Hochberg-adjusted P value; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-2.1 to 0.8]
Statistical Analysis 3: Comparison: B: GM-CSF + Attention Control Group vs D: Placebo + Attention Control Group; Test type: Superiority; p = 0.44, t-test, 2 sided — The P value is a Hochberg-adjusted P value; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.1 to 0.9]
Statistical Analysis 4: Comparison: C: Placebo + Supervised Exercise Therapy vs D: Placebo + Attention Control Group; Test type: Superiority; p < 0.01, t-test, 2 sided — The P value is a Hochberg-adjusted P value; Mean Difference (Final Values) = 3.7, 95% CI 2-sided [2.2 to 5.2]

4. Secondary Outcome: Change in CD34_CD45lo at 12-week Follow-up
Description: Red blood cells are lysed twice with freshly prepared lysis buffer. Remaining cells are stained with LIVE/DEAD® Fixable Dead Cell Stains for 20 minutes at room temperature and Fc receptors are blocked by incubating with Fc receptor blocking reagent for 10 minutes at 4oC. Samples are then stained with the following antibody cocktail for 30 minutes at 4oC: CD34 VioBlue, CD133-APC , CD45 AlexaFluor 700, and CD31 (PECAM-1) APC-eFluor® 780. Stained samples are acquired using a BD LSRII and analyzed using Flowjo software.
  The outcome is the absolute change in the percentages of cells.
Time Frame: change from baseline to week 12
Population: Note: It is pre-specified in the study protocol that investigators will determine whether a supervised treadmill exercise intervention alone (Group C) is associated with greater increases in CD34+ cells at 12-week follow-up, compared to Group D. Therefore, only group C and group D are included here.
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | C: Placebo + Supervised Exercise Therapy | D: Placebo + Attention Control Group
Number analyzed (Participants) | 48 | 43
percentage of cells | -0.002 [-0.006 to 0.003] | 0.004 [-0.001 to 0.008]
Statistical Analysis 1: Comparison: C: Placebo + Supervised Exercise Therapy vs D: Placebo + Attention Control Group; Test type: Superiority; p = 0.09, t-test, 2 sided; Mean Difference (Final Values) = -0.006, 95% CI 2-sided [-0.012 to 0.001]

5. Secondary Outcome: Change in CD34_CD45loCD133_ at 12-week Follow-up
Description: as for outcome 4
Time Frame: change from baseline to week 12
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | C: Placebo + Supervised Exercise Therapy | D: Placebo + Attention Control Group
Number analyzed (Participants) | 48 | 43
percentage of cells | -0.002 [-0.005 to 0.002] | 0.004 [0.000 to 0.007]
Statistical Analysis 1: Comparison: C: Placebo + Supervised Exercise Therapy vs D: Placebo + Attention Control Group; Test type: Superiority; p = 0.03, t-test, 2 sided; Mean Difference (Final Values) = -0.005, 95% CI 2-sided [-0.010 to -0.001]

6. Secondary Outcome: Change in CD34_CD45lo_CD31_ at 12-week Follow-up
Description: as for outcome 4
Time Frame: change from baseline to week 12
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | C: Placebo + Supervised Exercise Therapy | D: Placebo + Attention Control Group
Number analyzed (Participants) | 35 | 30
percentage of cells | -0.003 [-0.007 to 0.001] | 0.002 [-0.002 to 0.007]
Statistical Analysis 1: Comparison: C: Placebo + Supervised Exercise Therapy vs D: Placebo + Attention Control Group; Test type: Superiority; p = 0.09, t-test, 2 sided; Mean Difference (Final Values) = -0.005, 95% CI 2-sided [-0.012 to 0.001]

7. Secondary Outcome: Change in CD34_CD45lo_CD31_CD133_ at 12-week Follow-up
Description: as for outcome 4
Time Frame: change from baseline to week 12
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | C: Placebo + Supervised Exercise Therapy | D: Placebo + Attention Control Group
Number analyzed (Participants) | 35 | 30
percentage of cells | -0.003 [-0.006 to 0.001] | 0.001 [-0.003 to 0.005]
Statistical Analysis 1: Comparison: C: Placebo + Supervised Exercise Therapy vs D: Placebo + Attention Control Group; Test type: Superiority; p = 0.17, t-test, 2 sided; Mean Difference (Final Values) = -0.004, 95% CI 2-sided [-0.009 to 0.002]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected between randomization and final 26-week follow-up.
Arm/Group | A: GM-CSF + Supervised Treadmill Exercise Therapy | B: GM-CSF + Attention Control Group | C: Placebo + Supervised Exercise Therapy | D: Placebo + Attention Control Group
All-Cause Mortality (participants affected / at risk) | 2/53 | 1/53 | 0/53 | 0/51
Serious Adverse Events (participants affected / at risk) | 17/53 | 13/53 | 9/53 | 12/51
Other Adverse Events (participants affected / at risk) | 52/53 | 49/53 | 50/53 | 48/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: GM-CSF + Supervised Treadmill Exercise Therapy (N=53) | B: GM-CSF + Attention Control Group (N=53) | C: Placebo + Supervised Exercise Therapy (N=53) | D: Placebo + Attention Control Group (N=51)
Cardiovascular event (Cardiac disorders) | 4 (4) | 5 (6) | 2 (2) | 3 (3)
Diabetes (Endocrine disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General event (General disorders) | 7 (10) | 5 (5) | 4 (4) | 6 (6)
Infection (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular (Vascular disorders) | 2 (2) | 1 (1) | 2 (3) | 2 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: GM-CSF + Supervised Treadmill Exercise Therapy (N=53) | B: GM-CSF + Attention Control Group (N=53) | C: Placebo + Supervised Exercise Therapy (N=53) | D: Placebo + Attention Control Group (N=51)
Aching or soreness in feet (Musculoskeletal and connective tissue disorders) | 38 (126) | 36 (103) | 29 (100) | 22 (61)
Aching or soreness in thighs (Musculoskeletal and connective tissue disorders) | 27 (74) | 27 (53) | 26 (92) | 21 (53)
Aching or soreness in lower back (Musculoskeletal and connective tissue disorders) | 34 (120) | 37 (115) | 32 (136) | 32 (98)
Aching or soreness in knee joints (Musculoskeletal and connective tissue disorders) | 27 (82) | 26 (64) | 33 (120) | 22 (83)
Aching or soreness in other joints (Musculoskeletal and connective tissue disorders) | 14 (32) | 17 (37) | 16 (43) | 12 (25)
Aching or soreness in calves (Vascular disorders) | 40 (118) | 35 (86) | 36 (128) | 26 (70)
Aching or soreness in buttocks (Vascular disorders) | 25 (72) | 23 (53) | 22 (63) | 14 (34)
Aching or soreness in other areas (Musculoskeletal and connective tissue disorders) | 31 (68) | 30 (66) | 28 (61) | 21 (33)
Aching or soreness in hip joints (Musculoskeletal and connective tissue disorders) | 23 (59) | 23 (63) | 27 (93) | 21 (63)
Increase in shortness of breath (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 12 (20) | 8 (9) | 11 (14)
New chest pain (General disorders) | 4 (9) | 5 (6) | 3 (3) | 3 (4)
Fever greater than 101 degrees (General disorders) | 3 (3) | 3 (4) | 2 (2) | 3 (3)
Chills (General disorders) | 12 (26) | 22 (43) | 15 (29) | 12 (21)
New headaches (General disorders) | 25 (57) | 24 (40) | 19 (29) | 20 (39)
Pain in muscles (Musculoskeletal and connective tissue disorders) | 40 (109) | 38 (90) | 31 (103) | 28 (88)
Nausea or vomiting (Gastrointestinal disorders) | 13 (16) | 17 (27) | 17 (32) | 12 (19)
New rash (General disorders) | 11 (16) | 11 (15) | 10 (12) | 7 (12)
New swelling in hands or feet (General disorders) | 18 (28) | 18 (27) | 17 (23) | 16 (23)
Pain in bones (Musculoskeletal and connective tissue disorders) | 20 (38) | 19 (39) | 19 (30) | 17 (36)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other type of blood clotting or thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT01408901/Prot_SAP_000.pdf